CLINICAL TRIAL: NCT03249935
Title: Treatment Failure and Associated Predictors Following Azithromycin Treatment for Urogenital Chlamydial Infection in Males in Youth Correctional Facilities
Brief Title: YCFM (Youth Correctional Facilities Males)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0002; HHSN272201300012I
Record Dates: First submitted 2017-08-03; First posted 2017-08-15 (Actual); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-09

CONDITIONS: Chlamydial Infection
Keywords: Azithromycin; Chlamydia; Correctional; Facilities; Symptoms; Urethral; Urogenital; Youth
MeSH Terms: conditions — Chlamydia Infections | interventions — Azithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azithromycin (Experimental): Azithromycin 1 gm PO single dose given as directly observed
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 1 gm PO single dose given as directly observed

SUMMARY:
The proposed study is a single center (with multiple long-term YCFs) treatment trial of the CDC-recommended azithromycin regimen (1 gm PO once) for chlamydia in males. This study is designed primarily to determine the frequency of chlamydia treatment failure following azithromycin in males who do versus do not have urethral symptoms of urethral discharge and/or dysuria. Anticipated enrollment is 446 males, between the age of 12 to 21 years old, with subject participation duration of 28 days and study duration of 4 years. The primary objective of the study is to assess the microbiological efficacy of azithromycin in uncomplicated Chlamydia trachomatis infection in males with versus without urethral symptoms in YCFs.

DETAILED DESCRIPTION:
The proposed study is a single center (with multiple long-term YCFs) treatment trial of the CDC-recommended azithromycin regimen (1 gm PO once) for chlamydia in males residing in long-term gender-segregated YCFs. This study is designed primarily to determine the frequency of chlamydia treatment failure following azithromycin in males who do versus do not have urethral symptoms of urethral discharge and/or dysuria. Males age 12 to 21 years in good health (based on vital signs and provider's clinical evaluation documented in medical records) who are residing in long-term gender-segregated (not co-ed) YCFs (usual stay > 3 weeks) and who are identified as chlamydia-infected comprise the study population. The anticipated enrollment is 446 males with subject participation duration of 28 days and study duration of 4 years. The primary objective of the study is to assess the microbiological efficacy of azithromycin in uncomplicated Chlamydia trachomatis infection in males with versus without urethral symptoms in YCFs; in essence, this study will assess the frequency of chlamydia treatment failure to azithromycin at the Day 28 follow-up visit (Visit 2) in males with urethral symptoms compared to males without urethral symptoms. The secondary objective is to evaluate the association of laboratory findings (enrollment chlamydia load and OmpA genotype) and other participant characteristics (demographics, sexual behaviors, etc.) to chlamydia treatment failure in males after azithromycin treatment.

ELIGIBILITY:
Inclusion Criteria:

1.Male between the ages of 12 and 21 years 2.Residing in a long-term gender-segregated (no co-ed) YCF 3.Diagnosed with urogenital chlamydia as determined by a screening C. trachomatis NAAT 4.Anticipated length of stay at the YCF at the time of enrollment is at least 28 days 5.Willingness to provide written consent 6.Willingness to comply with study procedures

Exclusion Criteria:

1.Diagnosed with gonorrhea as determined by a screening Neisseria gonorrhoeae NAAT 2.Clinical diagnosis of epididymitis based on review of medical records 3.Known allergy to azithromycin, erythromycin, any macrolide or ketolide drug 4.History of liver problems due to use of azithromycin 5.Having received antimicrobial therapy with activity against C. trachomatis within 21 days of the positive chlamydia screening NAAT or in the interval between the positive screening NAAT and study enrollment 6.Any concomitant infection, which requires antimicrobial therapy with activity against C. trachomatis 7.Previously enrolled in this study 8.Unable to swallow pills 9.Other exclusion criteria, per clinician judgment, that prohibits subject from enrolling in study

Ages: 12 Years to 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County Department of Health Services - Juvenile Court Health Services, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin
Started | 100
Completed | 55
Not Completed | 45
Not completed — Discharged from facility early | 36
Not completed — Negative for chlamydia at enrollment | 4
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants who tested positive for chlamydia at baseline.
Arm/Group | Azithromycin
Number analyzed (Participants) | 96
Age, Continuous [Median (Full Range); unit: years] | 17.0 [15.2 to 18.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 38
  White | 11
  Other | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Experiencing Treatment Failure After Treatment With Azithromycin for Uncomplicated Chlamydia Trachomatis (CT) in Males With and Without Urethral Symptoms
Description: Test positive for Chlamydia trachomatis with Aptima Combo 2® Assay (AC2) and having enrollment and follow-up CT strains that had concordant genotyping of the CT major outer membrane protein (ompA) sequences or, if genotyping was unsuccessful on urine from both visits (i.e., due to insufficient number of ompA copies), then participants could not have unsupervised furloughs or report interim sex to be categorized as a treatment failure.
Time Frame: Day 28-follow-up visit
Population: Per protocol population, which included all participants who tested positive for CT at enrollment and were evaluable at day 28.
Measure: Count of Participants; unit: Participants
Groups:
- Symptomatic: Symptomatic was defined as urethral discharge and/or dysuria at baseline.
- Asymptomatic: Asymptomatic was defined as not having urethral discharge or dysuria at baseline.
Arm/Group | Symptomatic | Asymptomatic
Number analyzed (Participants) | 12 | 43
Participants | 1 | 3
Statistical Analysis 1: Comparison: Symptomatic vs Asymptomatic; Assumptions were that 20% of enrolled chlamydia-infected males will have urethral symptoms and azithromycin treatment failures will occur in 10% of symptomatic men vs. 2% of asymptomatic men. At a one-sided 0.05 significance level with power of 0.80, a sample size of 357 evaluable males would be needed, or approximately 72 symptomatic and 285 asymptomatic males. Assuming 20% of males enrolled would be unevaluable, a total of 446 males was targeted for enrollment; Test type: Superiority; Given that the study closed early and there were only 4 treatment failures, formal hypothesis testing was not performed

2. Secondary Outcome: Evaluate the Association of Laboratory Findings and Other Participant Characteristics to Chlamydia Treatment Failure in Males After Azithromycin Treatment
Description: Odds ratios for the outcome of treatment failure calculated for laboratory findings (enrollment chlamydia load and OmpA genotype) and other participant characteristics (demographics, sexual behaviors, etc.). Note that samples were not run for OmpA genotype.
Time Frame: Day 28-follow-up visit
Population: Per protocol population, which included all participants who tested positive for CT at enrollment and were evaluable for treatment failure at day 28.
Measure: Count of Participants; unit: Participants
Groups:
- Azithromycin: Azithromycin 1 gm PO single dose given as directly observed Azithromycin: Azithromycin 1 gm PO single dose given as directly observed
Arm/Group | Azithromycin
Number analyzed (Participants) | 55
Participants | 4
Statistical Analysis 1: Comparison: Azithromycin; Unadjusted odds ratio for age in years as a continuous variable in a logistic regression model predicting treatment failure at day 28; Test type: Superiority; p = 0.656, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.22 to 2.62]
Statistical Analysis 2: Comparison: Azithromycin; Unadjusted odds ratio for reporting at baseline new partners in the last 30 days (reference group=no new partners) from a logistic model predicting treatment failure at day 28; Test type: Superiority; p = 0.197, Regression, Logistic; Odds Ratio (OR) = 4.65, 95% CI 2-sided [0.45 to 47.89]
Statistical Analysis 3: Comparison: Azithromycin; Unadjusted odds ratio for Chlamydia viral load at baseline as a continuous variable in a logistic model predicting treatment failure at day 28; Test type: Superiority; p = 0.058, Regression, Logistic; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.45 to 1.01]

ADVERSE EVENTS:
Time Frame: After study drug administration (Study Visit 1) through the Day 28 follow-up visit (Study Visit 2).
Description: Gastrointestinal AEs that occur after study drug administration (Study Visit 1) and through the Day 28 follow-up visit (Study Visit 2) will be recorded. AEs which cause a participant to discontinue from the study after study drug administration (Study Visit 1) and through the Day 28 follow-up visit (Study Visit 2) will also be recorded.
Arm/Group | Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 5/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=100)
Nausea (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
In September 2018, the decision was made to stop enrollment early due to changes in the LA Public Health and YCF standard facility management systems; research staff were not able to overcome the resulting challenges making enrollment infeasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/35/NCT03249935/Prot_SAP_000.pdf